CLINICAL TRIAL: NCT06115525
Title: Isolated or Combined Use of NUTRIC Score and NRS-2002 to Predict Mortality in Patients Admitted to the Intensive Care Unit for Respiratory Failure
Brief Title: Isolated or Combined Use of NUTRIC Score and NRS-2002 to Predict Mortality in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Principal Investigator, Specialist Doctor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2627
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Nutrition Disorders; Malnutrition; Mortality
Keywords: mNUTRIC; NRS-2002; Respiratory Failure; Intensive Care Unit; Nutrition
MeSH Terms: conditions — Nutrition Disorders; Malnutrition; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Patients admitted to the intensive care unit due to respiratory failure with no mortality in the 3-month follow-up period
  Interventions: Other: mNUTRIC score; Other: NRS-2002
- Nonsurvivors: Patients who were admitted to the intensive care unit due to respiratory failure and mortality was observed in the 3-month follow-up period
  Interventions: Other: mNUTRIC score; Other: NRS-2002

INTERVENTIONS:
Other: mNUTRIC score — The mNUTRIC score is a useful means of gauging the nutritional risk of patients in intensive care. Originally designed for IC unit patients, the score is calculated even when patient cooperation is unfeasible, making it applicable for intubated patients. Information necessary for calculation can be obtained from the patient's kin. The mNUTRIC score (without IL-6) classifies patients according to predefined metrics. The following information is necessary: (1) the patient's age, (2) their APACHE II score, (3) their SOFA score, (4) their comorbidities, and (5) the number of days they were hospitalized before being admitted to ICU.
  Other Names: Modified Nutrition Risk in Critically Ill Score
Other: NRS-2002 — The NRS-2002 score is a tool utilised to measure the nutritional risk of patients in intensive care units. This tool was specifically developed for the purpose of evaluating intensive care unit patients and can be calculated without requiring the patient's active involvement. Additionally, it can be applied to patients who have been intubated and the required information can be sourced from their family members or relatives. The Nutritional Risk Screening (NRS)-2002 assesses a patient's nutritional risk based on five variables: (1) recent unexplained weight loss, (2) appetite, (3) BMI, (4) disease-related stress factors (comorbidities), and (5) age over 70 years which is an additional risk factor.
  Other Names: Nutritional Risk Score-2002

SUMMARY:
The objective of this investigation was to assess the predictive capacity of the NUTRIC Score and NRS-2002, separately or combined, in forecasting hospital, 28-day and 3-month mortality in patients with respiratory failure admitted to the intensive care unit.

DETAILED DESCRIPTION:
Malnutrition is a significant and widespread issue amongst hospitalized patients. Its prevalence is higher in critically ill patients who are admitted to Intensive Care Units (ICUs). Nutritional screening aims to estimate the probability of both positive and negative outcomes in patient treatment based on nutrition-related factors, and whether nutritional therapy can have a positive effect. The Nutritional Risk Score-2002 (NRS-2002) and Nutritional Risk Score in Critically Ill Patients (NUTRIC) are commonly used for nutritional risk assessment in critically ill patients. However, there is currently insufficient evidence in the literature to determine which scale should take precedence in the nutritional care protocol of critically ill patients with respiratory failure. Furthermore, there are no studies demonstrating the sensitivity of these scales varies based on the type of respiratory failure. This study aims to examine the effectiveness of the NUTRIC Score and NRS-2002, alone or combined, in predicting hospital, 28-day, and 3-month mortality in critically ill patients admitted to the intensive care unit with respiratory failure. Do the NUTRIC Score and NRS-2002 provide sufficient accuracy or is there a distinction when utilised singularly or together in forecasting mortality rates within the hospital, 28-day and 3-month time frames? Additionally, is there a defined threshold for predicting mortality in patients with respiratory failure when using the NUTRIC Score and NRS-2002 either by themselves or in conjunction? Does the efficacy of these prediction tools differ based on the type of respiratory failure?

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and over
* Admission to the intensive care unit due to respiratory failure (respiratory distress is included in the complaints of patients when admitted to the intensive care unit).

Exclusion Criteria:

* Patients diagnosed with neurodegenerative diseases (Alzheimer's disease and other dementia diseases, Parkinson's disease, Prion disease, Motor neuron diseases, Huntington's Disease, Spinocerebellar ataxia, Spinal muscular atrophy)
* Pregnant patients
* Patients with a length of stay in the ICU of less than 72 hours
* Patients in the terminal period who were diagnosed with malignancy and whose treatment process was terminated due to lack of response to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (aged ≥18) admitted to the Intensive Care Units at the Anesthesiology and Reanimation Clinic of Ankara Atatürk Sanatorium Training and Research Hospital with respiratory distress, who remain in ICU for over 72 hours and meet the study criteria, are included.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Mortality | 3 month
  Mortality data of patients admitted to the intensive care unit due to respiratory failure during 3-month follow-up period

SECONDARY OUTCOMES:
mNUTRIC score | 72 hours
  The mNUTRIC score is a useful means of gauging the nutritional risk of patients in intensive care. Originally designed for IC unit patients, the score is calculated even when patient cooperation is unfeasible, making it applicable for intubated patients. Information necessary for calculation can be obtained from the patient's kin. The mNUTRIC score (without IL-6) classifies patients according to predefined metrics. The following information is necessary: (1) the patient's age, (2) their APACHE II score, (3) their SOFA score, (4) their comorbidities, and (5) the number of days they were hospitalized before being admitted to ICU.
NRS-2002 score | 72 hours
  The NRS-2002 score is a tool utilised to measure the nutritional risk of patients in intensive care units. This tool was specifically developed for the purpose of evaluating intensive care unit patients and can be calculated without requiring the patient's active involvement. Additionally, it can be applied to patients who have been intubated and the required information can be sourced from their family members or relatives. The Nutritional Risk Screening (NRS)-2002 assesses a patient's nutritional risk based on five variables: (1) recent unexplained weight loss, (2) appetite, (3) BMI, (4) disease-related stress factors (comorbidities), and (5) age over 70 years which is an additional risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Onur KÜÇÜK, specialist, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No